CLINICAL TRIAL: NCT05397483
Title: Legal-Education Plus Trauma-informed Therapy to Improve Community Acceptance and Reintegration of Repentant Terrorists in Nigeria: A Pilot Randomised Controlled Trial
Brief Title: Legal-Education Plus Trauma-informed Therapy to Improve Community Acceptance and Reintegration of Repentant Terrorists in Nigeria
Acronym: LETiT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nottingham Trent University (Other)
Responsible Party: Principal Investigator, Dr Dung Jidong, PhD, Senior Lecturer, Nottingham Trent University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0000-0001-5034-0335d
Record Dates: First submitted 2022-05-25; First posted 2022-05-31 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Trauma, Psychological; Legal Education
MeSH Terms: conditions — Psychological Trauma | interventions — Methods

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LETiT (Experimental): The LETiT intervention will cover (a) Legal education with numerous aspects relating to human rights, access to legal support and tackling traumatic experiences.
  (b) The Trauma-informed Therapy component will involve addressing trauma, dispelling negative thoughts and building more positive thinking.
  It is worth adding that the LETiT intervention has undergone standardisation of procedure by adopting a coherent manual (e.g., the Legal Education plus Trauma-informed Therapy manual) specifically designed for the proposed intervention. For example, the legal education contents are collated from extant laws, including the 1999 Constitution of the Federal Republic of Nigeria.
  Interventions: Behavioral: Legal Education plus Trauma-informed Therapy (LETiT)
- Intervention As Usual (IAU) (Active Comparator): The Intervention As Usual (IAU) component of the proposed project is designed through a systematic collation of numerous government and non-governmental organisations' support information (e.g., news information and basic re-orientation of community members affected by terrorism). Thus, the IAU group will receive the government intervention involving media messages from the National Orientation Agency devoid of legal education or trauma-informed therapy.
  The training materials are organised to address key aspects of care such as (a) acknowledgement of the severity of lived experiences (b) reflection of current help received from the government and humanitarian services (c) essential aspects of self-care and caring for the vulnerable family and community members (d) inspiration for the future etc.
  Interventions: Behavioral: Intervention As Usual (IAU)

INTERVENTIONS:
Behavioral: Legal Education plus Trauma-informed Therapy (LETiT) — Group-1: Experimental (n=75 participants) will receive the LETiT which consists of a total of 12-group integrated sessions lasting approximately 60-90 minutes per session every week with 20-25 persons per sub-group.
  Arms: LETiT
Behavioral: Intervention As Usual (IAU) — Group-2: Controlled (n=75 participants) will receive the IAU which consists of a total of 12-group integrated sessions lasting approximately 60-90 minutes per session every week with 20-25 persons per sub-group.
  Arms: Intervention As Usual (IAU)

SUMMARY:
Terrorism is an issue of global concern, and reintegrating repentant terrorists, including their families, has often proved challenging considering the damages done by the terrorist group. Despite Boko Haram atrocities in Nigeria, the focus seems directed toward the repentant terrorists with limited attention to the communities, the trauma they suffered, and their involvement in the design of reintegration programmes. There is also limited community awareness of legal support channels to foster positive reintegration (Ike et al., 2021). The implication is that it risks undermining the social context that informs successful reintegration, improves acceptance, and reduces reoffending. However, there appears to be limited research on this important policy problem in Nigeria. Our study proposes to fill this gap by contributing to the research initiative through a novel cross-disciplinary intervention drawing on law and psychology entitled Legal Education plus Trauma-informed Therapy (LETiT) to improve community acceptance and reintegration of repentant terrorists in Nigeria.

ELIGIBILITY:
Inclusion Criteria:

* ages 18 - 85 years
* able to give consent
* able to understand and speak English
* score a minimum of 5 on Trauma Screening Questionnaire
* residents of designated communities of intervention (Adamawa, Maiduguri, and Plateau states)
* available for the study and follow up at 3- and 6-months post-intervention

Exclusion Criteria:

* less than 18 or above 85 years
* unable to give consent
* clinically diagnosed with severe PTSD/suicidal ideations or undergoing treatment
* temporary or non-residents who are unlikely to be available for follow up

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-06-20 (Estimated); Primary Completion 2023-06-19 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Trauma Screening Questionnaire | Change is being assessed at baseline, at 12 weeks end of intervention, at 3-months, and at 6-months post-intervention
  Change in traumatic experience is being assessed
Adaptive Stress Index | Change is being assessed at baseline, at 12 weeks end of intervention, at 3-months, and at 6-months post-intervention
  Change in stress is being assessed
Patient Health Questionnaire | Change is being assessed at baseline, at 12 weeks end of intervention, at 3-months, and at 6-months post-intervention
  Change in depression is being assessed
Generalised Anxiety Disorder Scale | Change is being assessed at baseline, at 12 weeks end of intervention, at 3-months, and at 6-months post-intervention
  Change in anxiety is being assessed
Legal-Education Awareness Scale | Change is being assessed at baseline, at 12 weeks end of intervention, at 3-months, and at 6-months post-intervention
  Change in awareness of human right is being assessed
Attitude Towards Repentant Terrorists and their Reintegration Scale | Change is being assessed at baseline, at 12 weeks end of intervention, at 3-months, and at 6-months post-intervention
  Change in of attitude towards repentant terrorists is being assessed
brief Verona Service Satisfaction Scale | Change is being assessed at 12 weeks end of intervention, at 3-months, and at 6-months post-intervention
  Change in service satisfaction is being assessed

CONTACTS AND LOCATIONS:
Overall Officials: Dung Jidong, PhD, Principal Investigator — Nottingham Trent University, UK

IPD SHARING:
Plan to Share IPD: Yes